CLINICAL TRIAL: NCT07294027
Title: Intracytoplasmic Sperm Injection (ICSI) Versus Conventional in Vitro Fertilization (IVF) in Couples With Unexplained Infertility: a Multicenter, Open-label, Parallel-group, Randomized Controlled Trial
Brief Title: ICSI Versus Conventional IVF in Couples With Unexplained Infertility
Acronym: ICSI/IVF-UI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Renmin Hospital of Wuhan University (Other); Jiaxing Maternity and Child Health Care Hospital (Other); Ningbo Women & Children's Hospital (Other); Beijing Obstetrics and Gynecology Hospital (Other); Xiangyang Central Hospital (Other); Huangshi Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-0689
Record Dates: First submitted 2025-08-27; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-08

CONDITIONS: Unexplained Infertility
Keywords: Unexplained infertility; Conventional in vitro fertilization; Intracytoplasmic sperm injection
MeSH Terms: interventions — Sperm Injections, Intracytoplasmic

STUDY DESIGN:
Intervention Model Description: This is a multicenter study. Each center enrolls participants using a competitive enrollment method and performs online randomization through the trial system. Using block randomization with a 1:1 allocation ratio, participants were assigned to either the ICSI group or the IVF group, with a block length set at 8. The trial system administrators were not involved in the treatment process. Eligible patients who provided informed consent were registered in the trial system by medical staff at each center on the day of oocyte retrieval. After entering participant information, the system automatically assigned patients based on pre-set parameters.
Masking Description: To safeguard patients' right to know and in accordance with previous similar studies, this study adopted an open-label design. Both participants and recruiters will be aware of the group assignments.
  However, the doctors performing embryo transfers, medical staff conducting routine prenatal check-ups and laboratory technicians analyzing biological samples will not be directly informed of whether patients participate in this clinical study and their grouping status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intracytoplasmic Sperm Injection (ICSI) (Active Comparator): All patients will receive controlled ovarian hyperstimulation (COH) treatment, which is performed by standard routines at each study center. The COH treatment includes either GnRH agonist protocol or GnRH antagonist protocol. Oocyte retrieval is scheduled for 36 (±2) hours after hCG injection. The retrieved cumulus oocyte complexes (COCs) will be allocated to undergo ICSI procedure according to the result of randomization.
  The first embryo transfer is performed using fresh embryo transfer (if without contraindication), limited to transferring 1-2 cleavage embryos or 1 blastocyst. The remaining available embryos will be frozen.
  Interventions: Procedure: ICSI
- Conventional in vitro fertilization (c-IVF) (Active Comparator): All patients will receive controlled ovarian hyperstimulation (COH) treatment, which is performed by standard routines at each study center. The COH treatment includes either GnRH agonist protocol or GnRH antagonist protocol. Oocyte retrieval is scheduled for 36 (±2) hours after hCG injection. The retrieved cumulus oocyte complexes (COCs) will be allocated to undergo conventional IVF procedure according to the result of randomization.
  The first embryo transfer is performed using fresh embryo transfer (if without contraindication), limited to transferring 1-2 cleavage embryos or 1 blastocyst. If the embryos in the IVF group are fertilized through different methods (some with late-RICSI), the first embryo transfer is limited to embryos fertilized through conventional IVF. The remaining available embryos will be frozen.
  Interventions: Procedure: IVF

INTERVENTIONS:
Procedure: ICSI — Insemination will be performed by using ICSI, 2 hours after oocyte retrieval. COCs will be stripped by using hyaluronidase. Only matured oocytes (MII stage) will be injected. Fertilization check will be performed at period of 16-18 hours after injection.
  Other standard assisted reproductive treatments are similar and parallel between two groups.
  Arms: Intracytoplasmic Sperm Injection (ICSI)
Procedure: IVF — Insemination will be performed by using conventional IVF, 2-4 hours after oocyte retrieval. Collected COCs will be inseminated (1-5×105 sperm/ml) and cultured overnight in culture medium. Fertilization check will be performed at period of 16-18 hours after insemination.
  If the IVF group experiences total fertilization failure or a fertilization rate of less than 25%, late rescue ICSI (Late-RICSI) will be performed on all MII stage oocytes using semen retained on the day of egg retrieval. The injection method is same as standard ICSI.
  Other standard assisted reproductive treatments are similar and parallel between two groups.
  Arms: Conventional in vitro fertilization (c-IVF)

SUMMARY:
This multicenter, open-label, parallel-group, randomized controlled trial aims to compare the live birth rate, fertilization outcomes, other pregnancy outcomes and safety between ICSI and conventional IVF among couples with unexplained infertility in China.

DETAILED DESCRIPTION:
A multicenter, large-scale, randomized controlled clinical trial will enroll 848 couples with unexplained infertility undergoing their first cycle of IVF or ICSI. The study will recruit participants from 6 Reproductive Medical Centers across mainland China. The participation in this study will be approximately 1 years with a total of 9 visits from controlled ovarian hyperstimulation, pregnancy to delivery. On the day of oocyte retrieval, eligible participants will be allocated to either the ICSI group or the IVF group in a 1:1 ratio. All participants will be randomized through block randomization, and each center will enroll participants using a competitive enrollment method.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 20-38 years
2. 18.5 < BMI < 24kg/m2
3. Couples diagnosed with primary unexplained infertility:

   * Regular menses or confirmed ovulation;

     * Normal ovarian reserve;

       * Patent fallopian tubes;

         * Normal uterus and cervix;

           * Normal endocrine profile;

             * Semen analysis meeting WHO 6th edition criteria

               * Normal karyotypes in both partners, no family history of genetic disorders
4. First IVF/ICSI cycle
5. Received GnRH agonist protocol or GnRH antagonist protocol
6. Willing to provide informed consent and comply with follow-up

Exclusion Criteria:

1. Preimplantation genetic testing (PGT) cycles
2. In vitro maturation (IVM) cycles
3. Using donor sperm/oocyte
4. Using frozen sperm/oocyte
5. <5 oocytes retrieved
6. Abnormal semen parameters on the day of oocyte retrieval
7. High risk of tubal pathology or endometriosis without laparoscopic exclusion
8. Untreated or poorly controlled endocrine disorders
9. Abnormal immune related examinations
10. Major organ/system disorders (cardiac, hepatic, renal, oncologic, hematologic, psychiatric, etc.)
11. Concurrent participation in other clinical trials.

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 848 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-07-30 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
Live birth rate after the first embryo transfer cycle | At birth
  Live birth is defined as the birth of at least one newborn after 24 weeks' gestation that exhibits any sign of life (twin will be a single count).

SECONDARY OUTCOMES:
Cumulative ongoing pregnancy rate within one year | At 12 weeks of gestation; At 12 months after randomization
  Achieving ongoing pregnancy within 12 months after randomization, regardless of the number of embryo transfers performed (limited to embryos obtained in the current study).
  Ongoing pregnancy refers to the presence of a gestational sac and fetal heart beat after 12 weeks of gestation.
Number of retrieved oocyte | 2 hours after oocyte retrieval
  Number of oocyte obtained on the day of oocyte retrieval
MII rate | 2 hours after oocyte retrieval
  [Only in ICSI group] The proportion of MII oocytes to the total number of retrieved oocytes.
Fertilization rate per oocyte inseminated/injected | At 16-18 hours after insemination or injection
  The proportion of fertilized oocytes to inseminated oocytes (IVF group) / injected oocytes (ICSI group).
Fertilization rate per oocyte retrieved | At 16-18 hours after insemination or injection
  The proportion of fertilized oocytes to the total number of retrieved oocytes.
Normal fertilization rate | At 16-18 hours after insemination or injection
  Normal fertilization is defined as the appearance of 2PN
Abnormal fertilization rate | At 16-18 hours after insemination or injection
  Abnormal fertilization is defined as the appearance of 1PN or ≥3PN
Degeneration rate of ICSI oocytes | At 16-18 hours after injection
  [Only in ICSI group] The proportion of oocytes that undergo degeneration assessed on Day 2 among all oocytes receiving ICSI.
Cleavage rate | At 16-18 hours after insemination or injection
  The proportion of normal cleavage observed on Day 2 in normally fertilized oocytes
Day 2 embryo formation rate | 2 days after oocyte retrieval
  The proportion of 4-cell stage embryos formed on Day 2 compared to normal fertilized oocytes.
Day 3 embryo formation rate | 3 days after oocyte retrieval
  The proportion of 8-cell stage embryos formed on Day 3 compared to normal fertilized oocytes.
Good quality embryo rate on Day 3 | 3 days after oocyte retrieval
  The proportion of I-II grade embryos with 6-10 cells on Day 3 compared to normal fertilized oocytes, according to Peter's scoring criteria.
Blastocyst formation rate | 6 days after oocyte retrieval
  The proportion of the number of blastocysts formed to the number of embryos undergoing blastocyst culture.
Good quality blastocyst formation rate | 6 days after oocyte retrieval
  The proportion of the number of blastocysts classified as 3BB or higher grade (according to Gardner scoring system) to the number of embryos undergoing blastocyst culture.
Good quality blastocyst rate | 6 days after oocyte retrieval
  The proportion of good quality blastocysts to the total number of blastocysts.
Number of available blastocyst | 6 days after oocyte retrieval
  Number of blastocysts of BC, CB grade and above, according to the Gardner scoring system.
Number of available embryo | 6 days after oocyte retrieval
  The total number of embryos that can be utilized for transplantation or cryopreservation.
Total fertilization failure rate | At 16-18 hours after insemination or injection
  Total fertilisation failure rate is defined as the absence of any zygotes with 2PN
Cycle cancellation rate | 6 days after oocyte retrieval
  The proportion of cycles with total fertilization failure or no available embryo to all oocyte retrieval cycles.
Moderate/severe ovarian hyperstimulation syndrome (OHSS) | At 10days after trigger; At 14 days after embryo transfer
  The exaggerated systemic response to ovarian stimulation. It is classified into mild, moderate, and severe based on the degree of bloating, ovarian volume enlargement, and respiratory, hemodynamic, and metabolic complications.
Positive pregnancy rate | 10-14 days after embryo transfer; At 12 months after randomization
  Positive pregnancy test is defined as a serum human chorionic gonadotropin level greater than 10mIU/mL after embryo transfer.
Clinical pregnancy rate | 30 days after embryo transfer
  Clinical pregnancy is defined as ultrasound detection of at least one gestational sac or other clear pregnancy manifestations under ultrasound (including clear ectopic pregnancy).
Implantation rate | 30 days after embryo transfer; At 12 months after randomization
  Implantation rate is defined as the number of gestational sacs per number of embryos transferred.
Ongoing pregnancy rate | At 12 weeks of gestation; At 12 months after randomization
  Ongoing pregnancy refers to the presence of a gestational sac and fetal heart beat after 12 weeks of gestation.
Ectopic pregnancy | 30 days after embryo transfer; At 12 months after randomization
  Ectopic pregnancy is defined as the presence of the gestational sac outside the uterine cavity detected by ultrasound.
Multiple pregnancy rate | 30 days after oocyte retrieval; At 12 months after randomization
  Multiple pregnancy is defined as the detection of two or more gestational sacs or positive heart beats by ultrasound.
Miscarriage rate | At 24 weeks of gestation; At 12 months after randomization
  Miscarriage refers to the loss of an intra-uterine pregnancy before 24 weeks of gestation.
Gestational diabetes mellitus | At 24-28 weeks of gestation
  Abnormal OGTT test
Hypertensive disorders of pregnancy | From 20 weeks of gestation up to at birth
  The hypertensive disorders of pregnancy include gestational hypertension, chronic hypertension, pre-eclampsia, chronic hypertension with preeclampsia, eclampsia and HELLP syndrome.
Antepartum haemorrhage | From 20 weeks of gestation up to at birth
  Vaginal bleeding caused by placenta previa, placental implantation, or unknown reasons in mid or late pregnancy.
Thrombotic diseases | From 20 weeks of gestation up to 4-6 weeks after birth
  If the participant experiences clinical symptoms such as lower limb pain, chest pain, hemoptysis, etc., and there is a high suspicion of thrombotic disease in clinical practice, confirmation will be made through examinations such as vascular ultrasound and CT angiography.
Gestational age at delivery | At birth
Preterm birth | At birth
  Pregnancy terminates after 28 weeks and before 37 weeks of gestation.
Spontaneous preterm birth | At birth
  Termination of pregnancy due to premature rupture of membranes or spontaneous uterine contractions between 28 to 37 weeks of gestation.
Iatrogenic preterm birth | At birth
  Termination of pregnancy due to iatrogenic factors between 28 to 37 weeks of gestation.
Birth weight | At birth
  Weight of newborn, classified as very low birth weight (<1500g), low birth weight (1500-2500g), macrosomia (>4000g).
Small for gestational age | At birth
  Birth weight below the 10th percentile for gestational age.
Large for gestational age | At birth
  Birth weight above the 90th percentile for gestational age.
Birth defect / Congenital anomaly | At birth; At 4-6 weeks after birth
  Any birth defect or congenital anomaly will be included.
NICU admission | At 4-6 weeks after birth
  The admittance of the newborn to NICU.
Perinatal mortality | At 4-6 weeks after birth
  Fetal or neonatal death occurring after 28 weeks of gestation, during delivery, or within 7 days after birth.
Neonatal mortality | At 4-6 weeks after birth
  Death of a live born baby within 28 days of birth.

CONTACTS AND LOCATIONS:
Overall Officials: Min Jin, PhD, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (7):
- China (7):
  - Beijing Obstetrics and Gynecology Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Huangshi Central Hospital, Huangshi, Hubei
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - Xiangyang Central Hospital, Xiangyang, Hubei
  - Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - Jiaxing Maternity and Child Health Care Hospital, Jiaxing, Zhejiang
  - Ningbo Women & Children's Hospital, Ningbo, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided